CLINICAL TRIAL: NCT01794481
Title: Benefits of Resistance Exercise Training in Locally Advanced Head and Neck Cancer Patients Undergoing Organ-Preserving Definitive Therapy
Brief Title: Benefits of Exercise Training in Head and Neck Cancer Patients Undergoing Organ-Preserving Definitive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011.070; HUM 33897 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2013-02-14; First posted 2013-02-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Participants allocated to usual care will receive their usual treatment program which will include dietician counseling as needed. As part of standardized care, participants will not be encouraged to begin a new exercise program(patients needing physical therapy at time of enrollment will be excluded.
- Resistance Exercise Training (Experimental): If you are randomized to the resistance exercise training (RET) program, you will undergo up to three 1-hour training sessions per week for 7 weeks during radiation therapy.
  There will be up to 3 sessions per week lasting up to one hour, and will generally include a 10- minute warm-up, rest periods and 10 minute cool-down. The goal is to perform the exercises as tolerated in week 1 and increase intensity as the weeks progress. Weights will be added each week depending on your tolerance to them. Rest periods will be incorporated into the exercises as needed. The intensity and weights used will be customized to the individual. During the home program portion, you will be asked to keep a weekly log of your exercises and the trainer will call you weekly to go over the log and provide support. At week 11 the trainer will meet with you to go over your individualized program and review your technique.
  Interventions: Procedure: Resistance Exercise Training (RET)

INTERVENTIONS:
Procedure: Resistance Exercise Training (RET) — If you are randomized to the resistance exercise training (RET) program, you will undergo up to three 1-hour training sessions per week for 7 weeks during radiation therapy.
  There will be up to 3 sessions per week lasting up to one hour, and will generally include a 10- minute warm-up, rest periods and 10 minute cool-down. The goal is to perform the exercises as tolerated in week 1 and increase intensity as the weeks progress. Weights will be added each week depending on your tolerance to them. Rest periods will be incorporated into the exercises as needed. The intensity and weights used will be customized to the individual. During the home program portion, you will be asked to keep a weekly log of your exercises and the trainer will call you weekly to go over the log and provide support. At week 11 the trainer will meet with you to go over your individualized program and review your technique.
  Arms: Resistance Exercise Training

SUMMARY:
The purpose of this study is to evaluate the potential benefit of an individualized resistance exercise-training program during radiotherapy for patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
Patients with locally advanced head and neck cancer are treated with radiation therapy (with/without chemotherapy) to avoid large surgical procedures. However, definitive radiation treatments can cause side effects (like mouth sores, difficulty swallowing) that often cause weight loss. It has been shown that a significant percentage of the weight loss is due to loss of muscle mass. Resistance exercise training works to increase muscle strength and endurance by doing repetitive exercises with weights, weight machines, or resistance bands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Joint Committee on Cancer (AJCC) stage II-IV head and neck squamous cell carcinoma who are beginning first-line non-surgical treatment with radiotherapy (with or without chemotherapy or targeted agents), and who are capable of understanding and adhering to the protocol requirements.
* Patients must be willing to comply with the study procedures and visits

Exclusion Criteria:

* Active cardiopulmonary disease
* Substantial dementia (based on Folstein Mini Mental State Examination <24 out of 30)
* Acute medical conditions, such as acute flare-up of joint condition or infection
* Participants must not be actively receiving physical therapy, at time of enrollment, or actively exercising 2 or more hours a day, with the intent to continue that regimen
* Patients refusing a percutaneous endoscopic gastrotomy (PEG) Tube needed for nutrition, as determined necessary by treating physician
* Patients are actively being treated for another cancer at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The effect of resistance exercise training (RET) versus usual care (UC) on the preservation of lean body mass. | 14 weeks
  Lean body mass will be analyzed at baseline, 3, 5, and 7-weeks (representing the last week of cancer treatment and end of on-site RET), 11-weeks (first clinic follow-up) and 14-weeks (second clinic follow-up and end of home-based RET program) for patients on both arms of the study.

SECONDARY OUTCOMES:
The effect of resistance exercise training (RET) versus usual care (UC) on the preservation of muscle strength. | 14 weeks
  Upper and lower body strength will be analyzed at baseline, 3, 5, and 7-weeks (representing the last week of cancer treatment and end of on-site RET), 11-weeks (first clinic follow-up) and 14-weeks (second clinic follow-up and end of home-based RET program) for patients on both arms of the study.
The effect of resistance exercise training (RET) versus usual care (UC) on six minute walk distance | 14 weeks
  The distance walked in six minutes at baseline will be compared to the distance walked at 14 weeks for both groups. These finding will then be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - Veterans Affairs (VA) Ann Arbor Healthcare System, Ann Arbor, Michigan
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan